CLINICAL TRIAL: NCT03136198
Title: B-lines Lung Ultrasound Guided ED Management of Acute Heart Failure Pilot Trial
Acronym: BLUSHED-AHF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Inova Fairfax Hospital (Other); Vanderbilt University (Other); Case Western Reserve University (Other); Wayne State University (Other)
Responsible Party: Principal Investigator, PETER S PANG, Associate Professor, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1R34HL136986-01 (NIH)
Record Dates: First submitted 2017-04-19; First posted 2017-05-02 (Actual); Results first posted 2020-05-20 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Heart Failure; Heart Failure Acute; Acute Cardiac Pulmonary Edema; Acute Cardiac Failure
Keywords: Heart Failure; Acute Heart Failure; Pulmonary Edema; Lung ultrasound; Extra vascular lung water; B-lines
MeSH Terms: conditions — Heart Failure; Pulmonary Edema | interventions — Vasodilator Agents; Noninvasive Ventilation

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Masking Description: A central, independent, Core Lab will review all images.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- LUS-guided strategy-of-care (Experimental): Patients randomized to the LUS strategy of care arm will be treated according to protocol. This protocol only involves therapies used in everyday AHF clinical practice.
  Interventions: Other: LUS-guided strategy-of-care; Drug: Intravenous Loop Diuretic; Drug: Vasodilator; Device: Non invasive Ventilation (NIV)
- Usual care (Placebo Comparator): Patients randomized to the usual care arm will also undergo lung ultrasound assessments. However, these results will not be revealed to the care team. Patients will receive treatment per usual, standard care.
  Interventions: Other: Usual Care; Drug: Intravenous Loop Diuretic; Drug: Vasodilator; Device: Non invasive Ventilation (NIV)

INTERVENTIONS:
Other: LUS-guided strategy-of-care — For patients randomized to the strategy-of-care arm, the LUS guided protocol will be initiated and continued until there is a decrease in B-lines to ≤ 15 or 6 hours of care has been delivered, whichever comes first.
  Treatment protocol:
  1. IV furosemide (unless already given): 2x single oral dose if on chronic therapy or 20-40 mg if diuretic naive.
  2. Optional therapies: non-invasive ventilation, vasodilators (SL, topical, or IV)
  3. Reassessment every 2 hours
  Arms: LUS-guided strategy-of-care
Other: Usual Care — Patients will receive usual AHF care
  Arms: Usual care
Drug: Intravenous Loop Diuretic — IV loop diuretic
Drug: Vasodilator — IV, topical, or SL Vasodilator
Device: Non invasive Ventilation (NIV) — Face, mouth, or nasal mask applied to provide positive pressure ventilation

SUMMARY:
Nearly 80% of acute heart failure (AHF) patients admitted to the hospital are initially treated in the emergency department (ED). Once admitted, within 30 days post-discharge, 27% of patients are re-hospitalized or die. Attempts to improve outcomes with novel therapies have all failed. The evidence for existing AHF therapies are poor: No currently used AHF treatment is known to improve outcomes. ED treatment is largely the same today as 40 years ago. Congestion, such as difficulty breathing, weight gain, and leg swelling, is the primary reason why patients present to the hospital for AHF. Treating congestion is the cornerstone of AHF management. Yet half of all AHF patients leave the hospital inadequately decongested. The investigators propose a novel approach to aggressively decongest patients in the ED setting: lung ultrasound guided, protocol driven, AHF management. LUS B-lines are a measure of extra-vascular lung water (EVLW). In the setting of AHF, LUS B-lines are a measure of congestion. This simple, easily learned technique has excellent reliability and reproducibility. The investigators hypothesize that a strategy-of-care will outperform usual care. At the present time, usual care is largely empirical. This study will improve the evidence base for ED AHF management. This proposed pilot study, if successful, will lead to an outcome trial examining whether an ED AHF strategy-of-care increases days alive and out of the hospital for patients.

DETAILED DESCRIPTION:
The primary goal of the BLUSHED AHF pilot trial is to determine whether an early lung ultrasound (LUS) guided, protocol-driven ED AHF strategy-of-care leads to more rapid and sustained resolution of congestion, as measured by LUS B-lines. If the investigators are able to demonstrate this necessary and sufficient information - targeted strategy-of-care is more effective than usual care - they will apply for a follow on study to achieve the following aim.

Aim 1: To demonstrate the effectiveness of a targeted decongestion strategy - LUS guided, protocol-driven ED AHF management - will result in improved 30-day outcomes vs. usual care. This aim will be tested using a randomized, controlled, unblinded, pragmatic, multi-center, simple trial design.

The pilot trial may determine that ED management alone is insufficient to impact the outcome. Thus, the investigators may need to modify their subsequent trial design to include targeted therapy throughout hospitalization. However, the pilot study will demonstrate whether targeted therapy effectively reduces B-lines.

PUBLIC HEALTH IMPACT Over one million hospitalizations for AHF occur every year in the US. Within 30 days after hospitalization, over 25% of AHF patients will be dead or re-hospitalized.4 Up to 67% of patients will be re-hospitalized and 36% will be dead by one year. For patients aged 65 years and older, AHF is the most common and most expensive reason for hospitalization. Despite major reductions in morbidity and mortality for chronic HF, considerably less progress has been seen in AHF.

Congestion is the primary reason why AHF patients present to the ED seeking medical care. Congestion is manifest by signs and symptoms of heart failure (HF); dyspnea, orthopnea, edema, and weight gain. Yet, how to best assess, grade, and manage congestion is not well established.

Freedom from congestion is associated with improved outcomes; Yet many patients leave the hospital inadequately decongested. The absence of robust, reliable methods to assess congestion is a primary reason why it is not well-assessed. A recent consensus statement published in 2010 highlights this fact: "…no method to assess congestion…has been validated." The investigators would argue many ED AHF patients are poorly assessed prior to treatment. In addition, they are poorly re-assessed prior to hospitalization to gauge the success or failure of initial management. While physical exam is currently the cornerstone of congestion assessment, it lacks sensitivity and inter-rater reliability.

The investigators challenge the current paradigm of relying on insensitive methods of congestion to guide therapy. Furthermore, they argue the lack of a robust evidence base for ED management of congestion contributes to poor outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 21 years
* Presents with shortness of breath at rest or with minimal exertion
* Clinical diagnosis of AHF and presence of > 15 total bilateral B-lines distributed in at least 4 zones on initial LUS
* Hx of chronic HF and any one of the following:

  * Chest radiograph consistent with AHF
  * Jugular venous distension
  * Pulmonary rales on auscultation
  * Lower extremity edema

Exclusion Criteria:

* Chronic renal dysfunction, including end-stage renal disease (ESRD) or estimated glomerular filtration rate (eGFR) < 45ml//min/1.73m2.
* Shock of any kind. Any requirement for vasopressors or inotropes.
* Systolic blood pressure (SBP) < 100 or >175 mmHg
* Need for immediate intubation
* Acute Coronary Syndrome- Presentation consistent with myocardial ischemia AND either new ST-segment elevation/depression
* Fever >101.5 ºF or chest radiograph or clinical picture of pneumonia
* End stage HF: transplant list, ventricular assist device
* Anemia requiring transfusion
* Known interstitial lung disease
* Suspected acute lung injury or acute respiratory distress syndrome (ARDS)
* Pregnant or recently pregnant within the last 6 months

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2017-07-10 (Actual); Primary Completion 2019-03-20 (Actual); Study Completion 2019-06-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter S Pang, MD, Principal Investigator — Indiana University
Locations (6):
- United States (6):
  - Eskenazi Health, Indianapolis, Indiana
  - IU Health Methodist Hospital, Indianapolis, Indiana
  - Detroit Receiving Hospital, Detroit, Michigan
  - Case Western Reserve University, Cleveland, Ohio
  - Vanderbilt University, Nashville, Tennessee
  - INOVA Health System, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pang PS, Russell FM, Ehrman R, Ferre R, Gargani L, Levy PD, Noble V, Lane KA, Li X, Collins SP. Lung Ultrasound-Guided Emergency Department Management of Acute Heart Failure (BLUSHED-AHF): A Randomized Controlled Pilot Trial. JACC Heart Fail. 2021 Sep;9(9):638-648. doi: 10.1016/j.jchf.2021.05.008. Epub 2021 Jul 7. PMID 34246609
- [Derived] Russell FM, Ehrman RR, Ferre R, Gargani L, Noble V, Rupp J, Collins SP, Hunter B, Lane KA, Levy P, Li X, O'Connor C, Pang PS. Design and rationale of the B-lines lung ultrasound guided emergency department management of acute heart failure (BLUSHED-AHF) pilot trial. Heart Lung. 2019 May-Jun;48(3):186-192. doi: 10.1016/j.hrtlng.2018.10.027. Epub 2018 Nov 15. PMID 30448355

RESULTS

PARTICIPANT FLOW:
Groups:
- LUS-guided Strategy-of-care: Patients randomized to the lung ultrasound (LUS) strategy of care arm will be treated according to protocol. This protocol only involves therapies used in everyday AHF clinical practice.
  LUS-guided strategy-of-care: For patients randomized to the strategy-of-care arm, the LUS guided protocol will be initiated and continued until there is a decrease in B-lines to ≤ 15 or 6 hours of care has been delivered, whichever comes first.
  Treatment protocol:
  1. IV furosemide (unless already given): 2x single oral dose if on chronic therapy or 20-40 mg if diuretic naive.
  2. Optional therapies: non-invasive ventilation, vasodilators (SL, topical, or IV)
  3. Reassessment every 2 hours
  Intravenous Loop Diuretic: IV loop diuretic
  Vasodilator: IV, topical, or SL Vasodilator
  Non invasive Ventilation (NIV): Face, mouth, or nasal mask applied to provide positive pressure ventilation
Period: Overall Study
Arm/Group | LUS-guided Strategy-of-care | Usual Care
Started | 66 | 64
Completed | 66 | 64
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- LUS-guided Strategy-of-care: Patients randomized to the LUS strategy of care arm will be treated according to protocol. This protocol only involves therapies used in everyday AHF clinical practice.
  LUS-guided strategy-of-care: For patients randomized to the strategy-of-care arm, the LUS guided protocol will be initiated and continued until there is a decrease in B-lines to ≤ 15 or 6 hours of care has been delivered, whichever comes first.
  Treatment protocol:
  1. IV furosemide (unless already given): 2x single oral dose if on chronic therapy or 20-40 mg if diuretic naive.
  2. Optional therapies: non-invasive ventilation, vasodilators (SL, topical, or IV)
  3. Reassessment every 2 hours
  Intravenous Loop Diuretic: IV loop diuretic
  Vasodilator: IV, topical, or SL Vasodilator
  Non invasive Ventilation (NIV): Face, mouth, or nasal mask applied to provide positive pressure ventilation
- Total: Total of all reporting groups
Arm/Group | LUS-guided Strategy-of-care | Usual Care | Total
Number analyzed (Participants) | 66 | 64 | 130
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.8 (15.9) | 66.2 (12.2) | 65.0 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 18 | 37
  Male | 47 | 46 | 93
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 63 | 61 | 124
  Unknown or Not Reported | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 35 | 34 | 69
  White | 30 | 29 | 59
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 66 | 64 | 130

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With B-lines ≤ 15 at the Conclusion of ED AHF Management
Description: B-lines ≤ 15 at the conclusion of ED AHF management or maximum of 6 hours after enrollment, whichever comes first.
Time Frame: During the ED phase of management, usually no more than 6 hours
Population: Out of the 130 participants a total of 8 (5 in the LUS-guided strategy of care arm and 3 in the Usual care arm) had a recorded ED discharge time which was prior to the first LUS, leaving 61 participants in each arm to be analyzed for the primary outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | LUS-guided Strategy-of-care | Usual Care
Number analyzed (Participants) | 61 | 61
Participants | 7 | 10

2. Other Pre Specified Outcome: Total Days Alive and Out Of Hospital (DAOOH)
Description: Total days alive and out of hospital through 30 and 90 days post-discharge
Time Frame: Up through 90 days, with specific reporting of events through 30 and 90 days
Reporting Status: Not Posted

3. Other Pre Specified Outcome: Association of B-lines at Discharge and 30-day / 90-day Outcomes
Time Frame: Up through 90 days, with specific reporting of events through 30 and 90 days
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Change in Biomarkers From Presentation to Pre-discharge
Time Frame: From admission to pre-discharge from the hospital, on average 5 to 7 days.
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Time to Reach B-lines <15
Time Frame: Throughout hospitalization, on average 5-7 days
Reporting Status: Not Posted

6. Other Pre Specified Outcome: B Lines < 15 at 24 Hours and at Discharge
Time Frame: Through the first 24 hours and then prior to discharge, on average 5-7 days after admission
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Composite of 30-day and 90-day All-cause Mortality, Cardiovascular (CV) Re-hospitalizations, and CV Emergency Department (ED) Revisits.
Description: CV endpoints are defined according to the 2014 American College of Cardiology/American Heart Association (ACC/AHA) Key Data Elements and Definitions for Cardiovascular Endpoint Events.
Time Frame: Up through 90 days, with specific reporting of events through 30 and 90 days
Reporting Status: Not Posted

8. Other Pre Specified Outcome: All Cause Readmissions, All Cause ED Re-visits
Description: 30- day and 90-day
Time Frame: Up through 90 days, with specific reporting of events through 30 and 90 days
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Number of Participants With Physical Exam Findings of Heart Failure When Discharge is Compared to Baseline
Description: Physical exam includes body weight, peripheral edema, jugular venous distention, pulmonary and cardiac auscultation
Time Frame: From admission throughout hospitalization, usually 5-7 days.
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Count of Pharmacologic Therapies the Patient Received in the ED
Description: This is a description of which pharmacologic therapies the patient has received.
Time Frame: From admission throughout hospitalization, usually 5-7 days.
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Count of Pharmacologic and Device Therapies the Patient Received During Hospitalization
Description: This is a description of which pharmacologic and device therapies the patient has received.
Time Frame: From admission throughout hospitalization, usually 5-7 days.
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Comparison of LUS Interpretation Within and Between Trained Investigators as Well as the Core Lab
Description: Calculation of intra and inter-agreement between investigators and also the Core Lab to determine the reproducibility of LUS
Time Frame: From admission throughout hospitalization, usually 5-7 days.
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Association of Baseline, Discharge, and Change With 30 and 90 Day Outcomes
Time Frame: Up through 90 days, with specific reporting of events through 30 and 90 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 7 days from consent
Arm/Group | LUS-guided Strategy-of-care | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/66 | 0/64
Serious Adverse Events (participants affected / at risk) | 2/66 | 2/64
Other Adverse Events (participants affected / at risk) | 8/66 | 15/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LUS-guided Strategy-of-care (N=66) | Usual Care (N=64)
NSTEMI (Cardiac disorders) | 1 (1) | 1 (1)
Gross hematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Mitral Regurgitation, severe (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LUS-guided Strategy-of-care (N=66) | Usual Care (N=64)
NSTEMI type 2 (Cardiac disorders) | 0 (0) | 5 (5)
Iron deficiency anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
MGUS, new diagnosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) — Subject was re-admitted due to abdominal pain caused by constipation
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 4 (4) | 4 (4)
Hyponatremia (Renal and urinary disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Hypotension (Renal and urinary disorders) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Vascular disorders) | 0 (0) | 1 (1) — Deep vein thrombosis and pulmonary embolism
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Hyponatremia (Cardiac disorders) | 1 (1) | 0 (0)
Cough (Cardiac disorders) | 1 (1) | 0 (0)
Supratherapeutic digoxin level (Cardiac disorders) | 1 (1) | 0 (0)
Nonsustained ventricular tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Mural thrombus (Cardiac disorders) | 0 (0) | 1 (1)
Mitral valve disease (Cardiac disorders) | 0 (0) | 1 (1)
Hypotension (Cardiac disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) — Asymptomatic

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-01-23): https://cdn.clinicaltrials.gov/large-docs/98/NCT03136198/Prot_SAP_002.pdf
  • Informed Consent Form (2018-11-08): https://cdn.clinicaltrials.gov/large-docs/98/NCT03136198/ICF_000.pdf